CLINICAL TRIAL: NCT01781819
Title: Ultrasound Based Acoustic Radiation Force Impulse (ARFI)Shear Wave Velocity Imaging (SVI)of the Kidneys in Pediatric Patients With Vesicoureteral Reflux
Brief Title: (ARFI) Shear Velocity Imaging of the Kidneys in Pediatric Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jonathan R. Dillman M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00063972
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Urine Reflux; Kidney Damage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARFI SVI ultrasound imaging (Experimental): Acoustic Radiation Force Impulse (ARFI) Shear Wave Velocity Imaging (SVI) ultrasound imaging
  Interventions: Procedure: ARFI SVI Ultrasound Imaging

INTERVENTIONS:
Procedure: ARFI SVI Ultrasound Imaging — Following a clinical renal ultrasound scan, the research scan using the ultrasound based acoustic radiation force impulse, or shear wave velocity imaging will be performed using standard approved ultrasound machines and transducers. This imaging will take approximately 5 to 10 minutes to complete.

SUMMARY:
Urine reflux (urine backing up into the kidneys) is common in the pediatric population and may be complicated by renal abnormalities, such as infection and scarring. Currently, urine reflux is detected using either voiding cystourethrogram or other procedures. A new technique called ultrasound-based Acoustic Radiation Force Impulse (ARFI), or shear wave velocity imaging SVI) is performed using standard approved ultrasound machines and transducers bu the sound waves/impulses are produced in a different pattern. We hope to evaluate the usefulness of ARFI in diagnosing possible kidney damage caused from urine reflux (urine backing up into the kidneys).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and younger
2. Are scheduled to have a clinically ordered kidney ultrasound and a voiding cystourethrogram (to evaluate urine reflux) on the same day. -

Exclusion Criteria:

None to list

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound-Based Acoustic Radiation Force Impulse(ARFI)Shear Wave Velocity Imaging (SVI) | 6 months
  To determine if this new ultrasound based imaging will effectively measure shear wave velocity in kidneys affected by urine reflux and be useful in determining the extent of kidney damage

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States